CLINICAL TRIAL: NCT00688376
Title: Randomized, Double-Blind, Placebo-Controlled Study of Efficacy and Safety of Donepezil Hydrochloride in Preadolescent and Adolescent Children With Attention Impairment Following Cancer Treatment
Brief Title: Efficacy and Safety of Donepezil Hydrochloride in Preadolescent and Adolescent Children With Attention Impairment Following Cancer Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-G000-333; E2020-G000-334 (Registry Identifier: NCT00687635); 2007-005435-28 (EudraCT Number); NCT00687635 (obsolete NCT alias)
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2015-11

CONDITIONS: Attention Impairment
Keywords: Attention; cancer; chemotherapy; donepezil; acetylcholinesterase; inhibitor
MeSH Terms: conditions — Neoplasms; Pain | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Donepezil hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil hydrochloride — During the 12-week Double-Blind Phase, subjects will receive oral donepezil hydrochloride tablets starting at a dose of 3 mg once daily. Doses will be increased incrementally at successive 3-week intervals on the basis of weight and tolerability. The final daily dose will be 3, 5, or 10 mg depending on body weight.
  During the Blinded Extension Phase, all subjects will receive active treatment (donepezil).
  Other Names: Aricept
  Arms: 1
Drug: Placebo — During the 12-week Double-Blind Phase, subjects will receive matching placebo tablets (3, 5, of 10 mg) once daily.
  During the 12-week Blinded Extension Phase, all subjects will receive active treatment (donepezil).
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of donepezil in children with persistent attention impairment that is present at least 12 months after the completion of cancer treatment.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, parallel group study in pediatric subjects who have persistent attention impairment following treatment for cancer. This trial has three phases: (1) pre-randomization to establish eligibility, (2) a 12-week, double-blind, placebo-controlled, parallel-group phase with dose escalation based on body weight, (3) a 12-week, blinded extension phase during which all subjects will receive active drug.

ELIGIBILITY:
1. The subject must have received at least one cycle of chemotherapy and/or cranial radiation, and must have completed this treatment at least one year before screening takes place for entry into this study.
2. Subjects may be male or female; age range: 6 - 17.5 years; weight ≥ 20 kg. They must be physically healthy and able to move about, with or without aids, must be living in the community, and must have adequate motor skills as shown by tests that will be given at the time of screening. The subject's eyesight and hearing must be good enough to allow cooperation with tests and physical examinations. Additionally, they must be able to swallow tablets.
3. There must be subjective complaints by subject and/or parent of difficulties in school or other daily activities, possibly related to impairments in attention. These difficulties must have emerged after treatment for cancer and must still be present 12 months after cessation of treatment. There must also be objective evidence for this impairment, as shown by a test that will be given to the subject at the time of screening.
4. The IQ must be >70 according to tests that will be given at the time of screening.
5. The first language in which the subject learned to read and write must be one that uses Roman lettering (a, b, c, etc.) and Arabic numerals (1, 2, 3, etc.).
6. The subject must not have previously taken any drugs in the class known as cholinesterase inhibitors.
7. A parent or legal guardian must be available who is willing and able to complete all of the outcome measures, to administer medications, and to accompany the subject to the required clinic visits.
8. Subjects with diabetes or thyroid disease may still be eligible if certain medical requirements are satisfied.
9. Female subjects who could become pregnant must undergo pregnancy testing and must agree to use contraception.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Inability to perform the required tests (for example, because of aphasia, motor deficits affecting the dominant hand, or mental retardation).
2. Motor coordination not sufficient, according to tests to be conducted at the time of screening.
3. Recurrence of cancer. If this happens, the subject will have to withdraw from the study.
4. Mental retardation/developmental disability.
5. Certain medications, such as methylphenidate, are not allowed during the study.
6. Major depression.
7. Problems with the digestive tract that could affect the subject's ability to absorb the study drug.
8. Hypersensitivity to a chemical class known as piperidine derivatives.
9. Certain other medical conditions as determined by clinical staff.
10. Alcoholism, drug abuse, or organic brain disease other than that caused by the cancer or its treatment.
11. Pregnancy, nursing, or unwillingness to undergo pregnancy testing if requested by clinical staff.
12. Pregnancy, lactation or plans to become pregnant, or unwilling to take a screening Beta-human chorionic gonadotropin (ßhCG) test if a female >10 years of age.
13. If sexually active, unwillingness to use birth control (males and females).
14. Plans for certain types of elective surgery that would occur while the study is in progress.
15. Plans for travel or other events that would interfere with the study schedule.
16. Active treatment with another investigational drug within 3 months of the screening visit.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2008-07-02 (Actual); Primary Completion 2009-05-26 (Actual); Study Completion 2009-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (13):
  - Stanford, California
  - Miami, Florida
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - Brooklyn, New York
  - Great Neck, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Oklahoma City, Oklahoma
  - Dallas, Texas
  - Houston, Texas
  - Road Runner Research Ltd., San Antonio, Texas
- Argentina (2):
  - Cordoba Capital, Córdoba Province
  - Buenos Aires
- Australia (2):
  - Sydney, New South Wales
  - Westmead, Sydney, New South Wales
- Calgary, Alberta, Canada
- Chile (2):
  - Antonio Varas, Providencia Santiago
  - Santa María, Providencia Santiago
- France (2):
  - Vandoeurvre Les Nancy
  - Villejuif
- Cologne, Germany
- Netherlands (4):
  - Amsterdam
  - Groningen
  - Rotterdam
  - Utrecht
- Spain (2):
  - Palma de Mallorca
  - Valencia
- Sutton, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 22 centers in the United States, France, Germany, the Netherlands, Spain, the UK, Argentina, Chile, and Australia during the period of 02 July 2008 to 26 May 2009.
Pre-assignment Details: This trial had three phases: (1)pre-randomization to establish eligibility; (2) a 12-week, double-blind, placebo-controlled, parallel-group phase with dose escalation based on body weight; (3) a 12-week, blinded extension phase during which all participants received active drug. Eligible participants were randomized to receive placebo or donepezil.
Groups:
- Donepezil: Donepezil 3 mg, 5 mg, or 10 mg donepezil Immediate Release (IR) orally, once daily
- Placebo: Placebo, matching 3 mg, 5 mg, and 10 mg placebo tablets administered orally, once daily
Period: Double-Blind Phase
Arm/Group | Donepezil | Placebo
Started | 40 | 32
Safety Population | 40 | 31
Completed | 34 | 25
Not Completed | 6 | 7
Not completed — Adverse Event | 4 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not treated | 0 | 1
Period: Blinded Extension Phase
Arm/Group | Donepezil | Placebo
Started | 34 | 25
Completed | 29 | 20
Not Completed | 5 | 5
Not completed — Adverse Event | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population (SP) included randomized participants who took at least one dose of study medication and who had at least one post-Baseline safety assessment. One participant from the placebo group was not evaluable for safety resulting in one less total participants (71) in the SP as compared to the randomized population (72).
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 40 | 31 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.1 (3.06) | 11.6 (2.83) | 11.9 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 25 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Test of Variables in Attention-Continuous Performance Test (TOVA-CPT) "D-prime" Standard Score (SS) at Week 12
Description: TOVA-CPT test has a standardized computer game-like format that tests attention and simple impulse control. It precisely measures a person's reaction time to clicking on correct targets versus incorrect targets. Scores are based on the number of "Hits" (correct responses), omission errors (failure to respond), commission errors/"False Alarms" (incorrect responses), response time, and sensitivity ("d-prime"). "D-prime" a dimensionless statistics is a measure of distractibility and reflects how well a person reacts correctly versus incorrectly. A higher value of "d-prime" is reached by having more "Hits" (correct response) and fewer "False Alarms" (incorrect response). Analysis was based on three factors: the "d-prime" standard score, reaction time variability standard score, and response time standard score. Standard scores less than or equal to 80 were significant for an attention deficit disorder. Standard scores greater than 80 were not significant for an attention deficit disorder.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Last Observed Carried Forward (LOCF) population included all safety participants for whom the TOVA-CPT "d-prime" standard score was available at both Screening and at least one "d-prime" score from the treatment period, in addition to having a post-Baseline safety assessment.
Measure: Mean (Standard Deviation); unit: d-prime
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 39 | 30
d-prime | 5.2 (8.77) | 4.5 (7.39)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; P-values, least squares (LS) mean, and 95% confidence interval (CI) were obtained from Analysis of Covariance (ANCOVA) model with treatment group as a factor and Baseline value as covariate; Test type: Superiority or Other; p = 0.694, ANCOVA; LS mean difference = 0.8, 95% CI 2-sided [-3.22 to 4.8]

2. Secondary Outcome: Change From Baseline in the TOVA-CPT "D-prime" Standard Score (SS) at Week 6
Description: as for outcome 1
Time Frame: Baseline and Week 6
Population: Intent-to-Treat (ITT) Last Observed Carried Forward (LOCF) population included all safety participants for whom the TOVA-CPT d-prime standard score was available at both Screening and at least one visit after the first dose of study drug during the Double-Blind Phase.
Measure: Mean (Standard Deviation); unit: d-prime
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 39 | 30
d-prime | 5.7 (8.41) | 6.2 (9.49)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.9458, ANCOVA; LS mean difference = -0.1, 95% CI 2-sided [-4.38 to 4.09]

3. Secondary Outcome: Change From Baseline in the Reaction Time Variability Standard Score (RTVSS) and Response Time Standard Score (RTSS) at Weeks 6 and 12
Description: The Reaction Time Variability is defined as the time measurement of how consistently the switch is pressed. The Response Time is the measurement of how fast or slow information is processed and responded to by the participant. The testing process was as described in a previous outcome measure. Standard scores less than or equal to 80 were significant for an attention deficit disorder. Standard scores greater than 80 were not significant for an attention deficit disorder.
Time Frame: Baseline, Weeks 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 39 | 30
milliseconds
  RTVSS (Week 6) | -3.4 (18.44) | -3.2 (15.75)
  RTVSS (Week 12) | -3.9 (15.21) | -5.0 (17.00)
  RTSS (Week 6) | -6.9 (13.17) | -9.6 (13.25)
  RTSS (Week 12) | -9.0 (13.15) | -9.1 (12.79)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; RTVSS Change from Baseline to Week 6 (LOCF). P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.743, ANCOVA; LS mean difference = -1.4, 95% CI 2-sided [-9.56 to 6.85]
Statistical Analysis 2: Comparison: Donepezil vs Placebo; RTVSS Change from Baseline to Week 12 (LOCF). P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.9561, ANCOVA; LS mean difference = 0.2, 95% CI 2-sided [-7.42 to 7.84]
Statistical Analysis 3: Comparison: Donepezil vs Placebo; RTSS Change from Baseline to Week 6 (LOCF). P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.4385, ANCOVA; LS mean difference = 2.5, 95% CI 2-sided [-3.97 to 9.04]
Statistical Analysis 4: Comparison: Donepezil vs Placebo; RTSS Change from Baseline to Week 12 (LOCF). P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.9088, ANCOVA; LS mean difference = -0.4, 95% CI 2-sided [-6.74 to 6]

4. Secondary Outcome: Change From Baseline in the Global Executive Composite Score, Behavioral Regulation Index, Metacognition Index, and Working Memory Subscale
Description: Behavioral Rating Inventory of Executive Functioning test evaluates impairment of executive function(planning and organization),memory,and sustained attention in children aged 5-18 years with wide range of developmental and acquired neurological conditions.Survey assess parent/guardian's perception of their child's executive functioning in home and school environments,which relate to daily function(as judged by parent).Each survey contains 86 items scored as;1(behavior is never a problem),2(behavior is sometimes a problem),or 3(behavior is often a problem).Data was presented as t-scores(raw scale scores are used to generate t-scores)for Global Executive Composite Score(t-score range 72-216),Behavioral Regulation Index(t-score range 28-84;inhibit,shift,and emotional control),Metacognition Inde (t-score range 44-132;initiate,working memory,plan/organize,organization of materials, and monitor),and Working Memory Subscale(t-score range 35-90).Higher scores indicate decline in performance.
Time Frame: Baseline and Week 12
Population: ITT population LOCF
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 39 | 30
t-scores
  Global Executive Composite Score | -1.3 (6.73) | -3.8 (6.78)
  Behavioral Regulation Index | 0.8 (7.54) | -1.9 (6.91)
  Metacognition Index | -2.3 (7.29) | -4.9 (6.99)
  Working Memory Scale | -3.6 (7.45) | -3.3 (6.59)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Global Executive Composite Score Analysis. P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.2886, ANCOVA; LS mean difference = 1.7, 95% CI 2-sided [-1.5 to 4.96]
Statistical Analysis 2: Comparison: Donepezil vs Placebo; Behavioral Regulation Index Analysis. P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.2555, ANCOVA; LS mean difference = 2.1, 95% CI 2-sided [-1.54 to 5.69]
Statistical Analysis 3: Comparison: Donepezil vs Placebo; Metacognition Index Analysis. P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.3155, ANCOVA; LS mean difference = 1.7, 95% CI 2-sided [-1.63 to 4.99]
Statistical Analysis 4: Comparison: Donepezil vs Placebo; Working Memory Scale Analysis. P-values, LS mean, and 95% confidence intervals were obtained from ANCOVA model with treatment group as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.9075, ANCOVA; LS mean difference = -0.2, 95% CI 2-sided [-3.55 to 3.16]

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were collected from the time the participant signed the informed consent form up to 30 days after discontinuation, or approximately 203 days.
Description: Safety population included randomized participants who received at least one dose of study medication and who had at least one post-Baseline safety assessment. Treatment-emergent adverse events (TEAEs), defined as an adverse event that started/increased in severity on/after the first dose of study medication are presented in this section.
Groups:
- Donepezil Double-Blind Phase; Donepezil Blinded Extension Phase: Donepezil 3 mg, 5 mg, or 10 mg donepezil Immediate Release (IR) orally, once daily
- Placebo Double-Blind Phase; Placebo Blinded Extension Phase: Placebo, matching 3 mg, 5 mg, and 10 mg placebo tablets administered orally, once daily
Arm/Group | Donepezil Double-Blind Phase | Placebo Double-Blind Phase | Donepezil Blinded Extension Phase | Placebo Blinded Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/31 | 0/34 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/31 | 0/34 | 0/25
Other Adverse Events (participants affected / at risk) | 30/40 | 20/31 | 21/34 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Double-Blind Phase (N=40) | Placebo Double-Blind Phase (N=31) | Donepezil Blinded Extension Phase (N=34) | Placebo Blinded Extension Phase (N=25)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Double-Blind Phase (N=40) | Placebo Double-Blind Phase (N=31) | Donepezil Blinded Extension Phase (N=34) | Placebo Blinded Extension Phase (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Precocious puberty (Endocrine disorders) | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Tear discoloration (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 2 | 1 | 3
Stomach discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 3
Asthenia (General disorders) | 0 | 2 | 1 | 1
Chills (General disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 2 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Xerosis (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 2 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 4
Dizziness exertional (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 10 | 7 | 2 | 6
Hyperreflexia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Abnormal behavior (Psychiatric disorders) | 1 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Nervous system disorders) | 0 | 1 | 0 | 1
Attention deficit/Hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 1 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Limitations of the study, such as early termination leading to small numbers of participants analyzed and technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No